CLINICAL TRIAL: NCT01597193
Title: A PHASE 1 OPEN-LABEL, DOSE ESCALATION STUDY EVALUATING THE SAFETY, TOLERABILITY, AND PHARMACOKINETICS OF ENZALUTAMIDE (FORMERLY MDV3100) IN PATIENTS WITH INCURABLE BREAST CANCER
Brief Title: Safety Study of Enzalutamide (MDV3100) in Patients With Incurable Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Astellas Pharma Inc (Industry); Medivation LLC, a wholly owned subsidiary of Pfizer Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: MDV3100-08; C3431006 (Other: Alias Study Number)
Record Dates: First submitted 2012-05-09; First posted 2012-05-11 (Estimated); Results first posted 2019-05-08 (Actual); Last update posted 2019-05-08 (Actual); Status verified 2019-05

CONDITIONS: Breast Cancer
Keywords: enzalutamide; MDV3100; breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — enzalutamide; Anastrozole; exemestane; Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- enzalutamide (80-mg with increase to 160 mg) (Experimental): enzalutamide be provided as two or four 40-mg capsules by mouth daily
  Interventions: Drug: enzalutamide
- enzalutamide and anastrozole (Experimental): enzalutamide (160 mg) administered as four 40-mg capsules by mouth once daily in combination with anastrozole (1 mg) administered as one 1-mg tablet by mouth once daily.
  Interventions: Drug: anastrozole; Drug: enzalutamide
- enzalutamide and exemestane 25 mg (Experimental): enzalutamide (160 mg) administered as four 40-mg capsules by mouth once daily in combination with exemestane administered as one 25-mg tablet daily
  Interventions: Drug: exemestane; Drug: enzalutamide
- enzalutamide and exemestane 50 mg (Experimental): enzalutamide (160 mg) administered as four 40-mg capsules by mouth once daily in combination with exemestane administered as two 25-mg tablets daily
  Interventions: Drug: enzalutamide; Drug: exemestane
- enzalutamide and fulvestrant (Experimental): enzalutamide (160 mg) administered as four 40-mg capsules by mouth once daily in combination with fulvestrant (500 mg) administered as two 250-mg intramuscular injections every 28 days
  Interventions: Drug: fulvestrant; Drug: enzalutamide

INTERVENTIONS:
Drug: enzalutamide — 80 mg (2 capsules) or 160 mg (4 capsules) taken orally daily.
  Other Names: MDV3100, Xtandi
  Arms: enzalutamide (80-mg with increase to 160 mg)
Drug: anastrozole — 1 mg/day
  Other Names: Arimidex
  Arms: enzalutamide and anastrozole
Drug: exemestane — The exemestane dose is 25mg daily.
  Other Names: Aromasin
  Arms: enzalutamide and exemestane 25 mg
Drug: fulvestrant — 500 mg every 28 days
  Other Names: Faslodex
  Arms: enzalutamide and fulvestrant
Drug: enzalutamide — 160 mg (4 capsules) taken orally daily.
  Other Names: MDV3100; Xtandi
  Arms: enzalutamide and anastrozole; enzalutamide and exemestane 25 mg; enzalutamide and exemestane 50 mg; enzalutamide and fulvestrant
Drug: exemestane — The exemestane dose is 50 mg daily.
  Other Names: Aromasin
  Arms: enzalutamide and exemestane 50 mg

SUMMARY:
The purpose of this study is to determine the safety, tolerability and pharmacokinetics of enzalutamide alone and in combination with anastrozole, or exemestane, or fulvestrant in patients with incurable breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed breast cancer with accompanying pathology report;
* Submit unstained representative tumor specimen, either as a paraffin block (preferred) or ≥ 10 unstained slides
* Received at least 2 lines of systemic therapy in the advanced setting (for enzalutamide alone arm only);
* Eastern Cooperative Oncology Group performance (ECOG) status of 0 or 1;
* Estimated life expectancy of at least 3 months

Exclusion Criteria:

* Severe concurrent disease, infection, or comorbidity that, in the judgment of the Investigator, would make the patient inappropriate for enrollment;
* Pregnant or lactating;
* Known or suspected brain metastasis or leptomeningeal disease;
* History of another malignancy within the previous 5 years other than curatively treated in situ carcinomas;
* For patients who are enrolled to receive enzalutamide plus anastrozole or exemestane or fulvestrant must not have received tamoxifen or any medication known to be a potent CYP3A4 inducer or inhibitor.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 101 (Actual)
Dates: Start 2012-04-30 (Actual); Primary Completion 2015-12-15 (Actual); Study Completion 2018-01-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (15):
- United States (15):
  - ATTN-Research Pharmacist, Aurora, Colorado
  - University of Colorado Cancer Center, Aurora, Colorado
  - University of Colorado Hospital, Anschutz Outpatient Pavilion, Aurora, Colorado
  - Connecticut Multispecialty Group, Enfield, Connecticut
  - Florida Cancer Specialists, Sarasota, Florida
  - Karmanos Cancer Institute, Detroit, Michigan
  - The West Clinic, PC, Corinth, Mississippi
  - The West Clinic, Southaven, Mississippi
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center - IDS Pharmacy, New York, New York
  - Memorial Sloan Kettering Cancer Center - OPD Pharmacy, New York, New York
  - The West Clinic, Germantown, Tennessee
  - The West Clinic, Memphis, Tennessee
  - Tennessee Oncology, PLLC., Nashville, Tennessee
  - The Sarah Cannon Research Institute, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Stage 1: Included participants with incurable breast cancer. Stage 2: Included participants with hormone receptor-positive incurable breast cancer.
Groups:
- Dose Escalation: Enzalutamide 80 mg: Participants received enzalutamide 80 milligram (mg) (two 40 mg) capsules, orally, once daily until documented disease progression, initiation of a new antitumor treatment, an intolerable adverse event (including any seizure), noncompliance, withdrawal of consent, discontinuation by sponsor, or investigator. Participants were followed-up until 30 days after last dose of study drug or before initiation of a new antitumor or investigational therapy, whichever occurred first.
- Dose Escalation: Enzalutamide 160 mg: Participants received enzalutamide 160 mg (four 40 mg) capsules, orally, once daily until documented disease progression, initiation of a new antitumor treatment, an intolerable adverse event (including any seizure), noncompliance, withdrawal of consent, discontinuation by sponsor, or investigator. Participants were followed-up until 30 days after last dose of study drug or before initiation of a new antitumor or investigational therapy, whichever occurred first.
- Dose Expansion: Enzalutamide 160 mg: Participants received enzalutamide 160 mg (four 40 mg) capsules, orally, once daily until documented disease progression, initiation of a new antitumor treatment, an intolerable adverse event (including any seizure), noncompliance, withdrawal of consent, discontinuation by the sponsor, or investigator. Participants were followed-up until 30 days after last dose of study drug or before initiation of a new antitumor or investigational therapy, whichever occurred first.
- Dose Expansion: Enzalutamide 160 mg + Anastrozole 1 mg: Participants received enzalutamide 160 mg (four 40 mg) capsule in combination with the anastrozole 1 mg tablet, orally, once daily until documented disease progression, initiation of a new antitumor treatment, an intolerable adverse event (including any seizure), noncompliance, withdrawal of consent, discontinuation by sponsor, or investigator. Participants were followed-up until 30 days after last dose of study drug or before initiation of a new antitumor or investigational therapy, whichever occurred first.
- Dose Expansion: Enzalutamide 160 mg + Exemestane 25 mg: Participants received enzalutamide 160 mg (four 40 mg) capsule in combination with the exemestane 25 mg tablet, orally, once daily until documented disease progression, initiation of a new antitumor treatment, an intolerable adverse event (including any seizure), noncompliance, withdrawal of consent, discontinuation by sponsor, or investigator. Participants were followed-up until 30 days after last dose of study drug or before initiation of a new antitumor or investigational therapy, whichever occurred first.
- Dose Expansion: Enzalutamide 160 mg + Exemestane 50 mg: Participants received enzalutamide 160 mg (four 40 mg) capsule in combination with the exemestane 50 mg tablet, orally, once daily until documented disease progression, initiation of a new antitumor treatment, an intolerable adverse event (including any seizure), noncompliance, withdrawal of consent, discontinuation by sponsor, or investigator. Participants were followed-up until 30 days after last dose of study drug or before initiation of a new antitumor or investigational therapy, whichever occurred first.
- Dose Expansion: Enzalutamide 160 mg + Fulvestrant 500 mg: Participants received enzalutamide 160 mg (four 40 mg) capsule once daily in combination with the fulvestrant 500 mg intramuscular injection, once every 28 days until documented disease progression, initiation of a new antitumor treatment, an intolerable adverse event (including any seizure), noncompliance, withdrawal of consent, discontinuation by the sponsor, or investigator. Participants were followed-up until 30 days after last dose of study drug or before initiation of a new antitumor or investigational therapy, whichever occurred first.
Period: Stage 1: Dose Escalation (141 Days)
Arm/Group | Dose Escalation: Enzalutamide 80 mg | Dose Escalation: Enzalutamide 160 mg | Dose Expansion: Enzalutamide 160 mg | Dose Expansion: Enzalutamide 160 mg + Anastrozole 1 mg | Dose Expansion: Enzalutamide 160 mg + Exemestane 25 mg | Dose Expansion: Enzalutamide 160 mg + Exemestane 50 mg | Dose Expansion: Enzalutamide 160 mg + Fulvestrant 500 mg
Started | 7 | 8 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 7 | 8 | 0 | 0 | 0 | 0 | 0
Not completed — Disease progression | 7 | 8 | 0 | 0 | 0 | 0 | 0
Period: Stage 2: Dose Expansion (1067 Days)
Arm/Group | Dose Escalation: Enzalutamide 80 mg | Dose Escalation: Enzalutamide 160 mg | Dose Expansion: Enzalutamide 160 mg | Dose Expansion: Enzalutamide 160 mg + Anastrozole 1 mg | Dose Expansion: Enzalutamide 160 mg + Exemestane 25 mg | Dose Expansion: Enzalutamide 160 mg + Exemestane 50 mg | Dose Expansion: Enzalutamide 160 mg + Fulvestrant 500 mg
Started | 0 | 0 | 14 | 20 | 16 | 23 | 11
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 14 | 20 | 16 | 23 | 11
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 2 | 3 | 0
Not completed — Disease progression | 0 | 0 | 14 | 18 | 14 | 18 | 11
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis population included all enrolled participants who received at least 1 dose of Enzalutamide.
Groups:
- Dose Escalation: Enzalutamide 80 mg: Participants received enzalutamide 80 mg (two 40 mg) capsules, orally, once daily until documented disease progression, initiation of a new antitumor treatment, an intolerable adverse event (including any seizure), noncompliance, withdrawal of consent, discontinuation by sponsor, or investigator. Participants were followed-up until 30 days after last dose of study drug or before initiation of a new antitumor or investigational therapy, whichever occurred first.
- Total: Total of all reporting groups
Arm/Group | Dose Escalation: Enzalutamide 80 mg | Dose Escalation: Enzalutamide 160 mg | Dose Expansion: Enzalutamide 160 mg | Dose Expansion: Enzalutamide 160 mg + Anastrozole 1 mg | Dose Expansion: Enzalutamide 160 mg + Exemestane 25 mg | Dose Expansion: Enzalutamide 160 mg + Exemestane 50 mg | Dose Expansion: Enzalutamide 160 mg + Fulvestrant 500 mg | Total
Number analyzed (Participants) | 7 | 8 | 14 | 20 | 16 | 23 | 11 | 99
Age, Customized [Count of Participants; unit: Participants]
  Less than (<) 65 years | 6 | 5 | 11 | 12 | 13 | 10 | 6 | 63
  Between 65 to 74 years | 1 | 3 | 2 | 5 | 2 | 12 | 4 | 29
  Greater than or equal to (>=) 75 years | 0 | 0 | 1 | 3 | 1 | 1 | 1 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 14 | 20 | 16 | 23 | 11 | 99
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Dose-Escalation Phase: Percentage of Participants With Dose-limiting Toxicity (DLTs)
Description: DLTs were defined as any of following events related to the study drug: Any adverse event (AE) consistent with a seizure of any grade; Grade greater than equal to (>=) 3 fatigue, diarrhea, nausea, or vomiting that did not improve to Grade 1 within 14 days of initiating standard of care therapy; any Grade >=3 hematologic toxicity with the following modifications: 1) Grade >=3 platelet count associated with bleeding, 2) Grade >=3 absolute neutrophil count that persists for 7 or more days or that was associated with fevers (febrile neutropenia); Grade >=3 any other non-hematological toxicity that was determined to be related to study drug.
Time Frame: Baseline up to Day 35
Population: Safety analysis population included all enrolled participants who received at least 1 dose of Enzalutamide. Here, number of participants analyzed signifies those participants who were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Dose Escalation: Enzalutamide 80 mg | Dose Escalation: Enzalutamide 160 mg
Number analyzed (Participants) | 6 | 7
percentage of participants | 16.7 | 0.0

2. Primary Outcome: Percentage of Participants With Adverse Events of Grade 3 or Higher Severity by National Cancer Institute Common Toxicity Criteria For Adverse Events (NCI CTCAE) (Version 4.03)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. AE was assessed according to severity grading based on NCI CTCAE Version 4.03 and defined as Grade 3 AEs = severe or medically significant events but not immediately life-threatening, hospitalization or prolongation of hospitalization indicated, disabling, limiting self-care activities of daily living; Grade 4 AEs = life-threatening, urgent intervention indicated; Grade 5 AEs = death related to adverse event.
Time Frame: Day 1 up to 30 days after the last dose of study drug or before initiation of a new systemic antitumor treatment, whichever occurred first (up to 3.5 years)
Population: Safety analysis population included all enrolled participants who received at least 1 dose of Enzalutamide.
Measure: Number; unit: percentage of participants
Arm/Group | Dose Escalation: Enzalutamide 80 mg | Dose Escalation: Enzalutamide 160 mg | Dose Expansion: Enzalutamide 160 mg | Dose Expansion: Enzalutamide 160 mg + Anastrozole 1 mg | Dose Expansion: Enzalutamide 160 mg + Exemestane 25 mg | Dose Expansion: Enzalutamide 160 mg + Exemestane 50 mg | Dose Expansion: Enzalutamide 160 mg + Fulvestrant 500 mg
Number analyzed (Participants) | 7 | 8 | 14 | 20 | 16 | 23 | 11
percentage of participants | 57.1 | 12.5 | 21.4 | 30.0 | 37.5 | 39.1 | 36.4

3. Primary Outcome: Percentage of Participants With Treatment-Emergent Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study treatment without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death, initial or prolonged inpatient hospitalization, life-threatening experience (immediate risk of dying), persistent or significant disability or incapacity, congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 30 days after last dose of study drug that were absent before treatment or that worsened relative to pretreatment state. AEs included both serious and non-serious adverse events.
Time Frame: as for outcome 2
Population: Safety analysis population included all enrolled participants who received at least 1 dose of Enzalutamide.
Measure: Number; unit: percentage of participants
Arm/Group | Dose Escalation: Enzalutamide 80 mg | Dose Escalation: Enzalutamide 160 mg | Dose Expansion: Enzalutamide 160 mg | Dose Expansion: Enzalutamide 160 mg + Anastrozole 1 mg | Dose Expansion: Enzalutamide 160 mg + Exemestane 25 mg | Dose Expansion: Enzalutamide 160 mg + Exemestane 50 mg | Dose Expansion: Enzalutamide 160 mg + Fulvestrant 500 mg
Number analyzed (Participants) | 7 | 8 | 14 | 20 | 16 | 23 | 11
percentage of participants | 28.6 | 12.5 | 14.3 | 5.0 | 31.3 | 13.0 | 18.2

4. Primary Outcome: Percentage of Participants Who Discontinued the Study Drug Due to Adverse Events or Serious Adverse Events
Description: An AE was any untoward medical occurrence in a participant who received study treatment without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death, initial or prolonged inpatient hospitalization, life-threatening experience (immediate risk of dying), persistent or significant disability or incapacity, congenital anomaly.
Time Frame: as for outcome 2
Population: Safety analysis population included all enrolled participants who received at least 1 dose of Enzalutamide.
Measure: Number; unit: percentage of participants
Arm/Group | Dose Escalation: Enzalutamide 80 mg | Dose Escalation: Enzalutamide 160 mg | Dose Expansion: Enzalutamide 160 mg | Dose Expansion: Enzalutamide 160 mg + Anastrozole 1 mg | Dose Expansion: Enzalutamide 160 mg + Exemestane 25 mg | Dose Expansion: Enzalutamide 160 mg + Exemestane 50 mg | Dose Expansion: Enzalutamide 160 mg + Fulvestrant 500 mg
Number analyzed (Participants) | 7 | 8 | 14 | 20 | 16 | 23 | 11
percentage of participants | 0.0 | 0.0 | 7.1 | 5.0 | 12.5 | 13.0 | 0.0

5. Primary Outcome: Percentage of Participants Who Require Dose Reductions Due to Adverse Events
Description: as for outcome 4
Time Frame: as for outcome 2
Population: Safety analysis population included all enrolled participants who received at least 1 dose of Enzalutamide.
Measure: Number; unit: percentage of participants
Arm/Group | Dose Escalation: Enzalutamide 80 mg | Dose Escalation: Enzalutamide 160 mg | Dose Expansion: Enzalutamide 160 mg | Dose Expansion: Enzalutamide 160 mg + Anastrozole 1 mg | Dose Expansion: Enzalutamide 160 mg + Exemestane 25 mg | Dose Expansion: Enzalutamide 160 mg + Exemestane 50 mg | Dose Expansion: Enzalutamide 160 mg + Fulvestrant 500 mg
Number analyzed (Participants) | 7 | 8 | 14 | 20 | 16 | 23 | 11
percentage of participants | 0.0 | 0.0 | 0.0 | 20.0 | 12.5 | 8.7 | 18.2

6. Primary Outcome: Percentage of Participants With Potentially Clinically Significant Change From Baseline in Vital Signs
Description: Absolute systolic blood pressure (SBP) greater than (>) 180 millimeter of mercury (mm Hg) and an increase of >40 mm Hg from baseline; absolute SBP less than (<) 90 mm Hg and an decrease of >30 mm Hg from baseline. Absolute diastolic blood pressure (DBP) >105 mm Hg and an increase of >30 mm Hg from baseline; absolute DBP <50 mm Hg and an increase of >20 mm Hg from baseline. Absolute heart rate >120 beats per minute (bpm) and an increase of >30 bpm from baseline; absolute heart rate <50 bpm and decrease of >20 bpm from baseline. Participants with any of these abnormalities were reported for this outcome in each arm.
Time Frame: as for outcome 2
Population: Safety analysis population included all enrolled participants who received at least 1 dose of Enzalutamide.
Measure: Number; unit: percentage of participants
Arm/Group | Dose Escalation: Enzalutamide 80 mg | Dose Escalation: Enzalutamide 160 mg | Dose Expansion: Enzalutamide 160 mg | Dose Expansion: Enzalutamide 160 mg + Anastrozole 1 mg | Dose Expansion: Enzalutamide 160 mg + Exemestane 25 mg | Dose Expansion: Enzalutamide 160 mg + Exemestane 50 mg | Dose Expansion: Enzalutamide 160 mg + Fulvestrant 500 mg
Number analyzed (Participants) | 7 | 8 | 14 | 20 | 16 | 23 | 11
percentage of participants
  Blood pressure | 1 | 0 | 1 | 0 | 1 | 2 | 1
  Heart rate | 0 | 2 | 1 | 0 | 0 | 0 | 0

7. Primary Outcome: Dose-Escalation Phase: Maximum Plasma Concentration (Cmax) of Enzalutamide and Its Metabolites After Single Dose
Description: Carboxylic Acid (M1) and N-desmethyl (M2) are two metabolites of Enzalutamide.
Time Frame: pre-dose, 0.5, 1, 2, 4, 6, 24, 48, 72 and 96 hours post dose on Day 1
Population: Pharmacokinetic (PK) analysis population included all participants who had at least 1 dose of Enzalutamide and had sufficient PK data to calculate at least 1 of the PK parameters of interest in at least 1 treatment period.
Measure: Mean (Standard Deviation); unit: micrograms per milliliter
Arm/Group | Dose Escalation: Enzalutamide 80 mg | Dose Escalation: Enzalutamide 160 mg
Number analyzed (Participants) | 7 | 8
micrograms per milliliter
  Enzalutamide | 1.90 (0.757) | 4.01 (2.09)
  M1 | 0.0375 (0.0286) | 0.0707 (0.0379)
  M2 | 0.0879 (0.0718) | 0.184 (0.0689)

8. Primary Outcome: Dose-Escalation Phase: Time to Reach Maximum Plasma Concentration (Tmax) of Enzalutamide and Its Metabolites After Single Dosing
Description: Carboxylic Acid (M1) and N-desmethyl (M2) are two metabolites of Enzalutamide.
Time Frame: pre-dose, 0.5, 1, 2, 4, 6, 24, 48, 72 and 96 hours post dose on Day 1
Population: PK analysis population included all participants who had at least 1 dose of Enzalutamide and had sufficient PK data to calculate at least 1 of the PK parameters of interest in at least 1 treatment period.
Measure: Median (Full Range); unit: hours
Arm/Group | Dose Escalation: Enzalutamide 80 mg | Dose Escalation: Enzalutamide 160 mg
Number analyzed (Participants) | 7 | 8
hours
  Enzalutamide | 0.500 [0.500 to 2.00] | 1.00 [0.350 to 4.00]
  M1 | 24.1 [5.55 to 25.1] | 23.1 [4.00 to 23.9]
  M2 | 23.9 [21.1 to 25.1] | 23.7 [20.8 to 24.5]

9. Primary Outcome: Dose-Escalation Phase: Area Under the Plasma Concentration-time Curve From Time Zero to 24 Hours (AUC24h) of Enzalutamide and Its Metabolites After Single Dose
Description: Carboxylic Acid (M1) and N-desmethyl (M2) are two metabolites of Enzalutamide.
Time Frame: pre-dose, 0.5, 1, 2, 4, 6 and 24 hours post dose on Day 1
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: micrograms*hour per milliliter
Arm/Group | Dose Escalation: Enzalutamide 80 mg | Dose Escalation: Enzalutamide 160 mg
Number analyzed (Participants) | 7 | 8
micrograms*hour per milliliter
  Enzalutamide | 17.3 (8.32) | 41.6 (8.19)
  M1 | 0.632 (0.385) | 1.20 (0.648)
  M2 | 1.13 (0.916) | 2.76 (1.00)

10. Primary Outcome: Dose-Escalation Phase: Area Under the Plasma Concentration-time Curve From Time Zero to 72 Hours (AUC72h) of Enzalutamide After Single Dosing
Time Frame: pre-dose, 0.5, 1, 2, 4, 6, 24, 48 and 72 hours post dose on Day 1
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: micrograms*hour per milliliter
Arm/Group | Dose Escalation: Enzalutamide 80 mg | Dose Escalation: Enzalutamide 160 mg
Number analyzed (Participants) | 7 | 8
micrograms*hour per milliliter | 43.0 (21.4) | 107 (15.6)

11. Primary Outcome: Dose-Escalation Phase: Area Under the Plasma Concentration-Time Profile From Time Zero Extrapolated to Infinite Time (AUCinf) of Enzalutamide After Single Dosing
Description: AUCinf = Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - inf).
Time Frame: pre-dose, 0.5, 1, 2, 4, 6, 24, 48, 72 and 96 hours post dose on Day 1
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: micrograms*hour per milliliter
Arm/Group | Dose Escalation: Enzalutamide 80 mg | Dose Escalation: Enzalutamide 160 mg
Number analyzed (Participants) | 7 | 8
micrograms*hour per milliliter | 208 (66.0) | 478 (232)

12. Primary Outcome: Dose-Escalation Phase: Terminal Elimination Half-Life (t1/2) of Enzalutamide After Single Dosing
Description: Terminal elimination half-life is the time measured for the plasma concentration of Enzalutamide to decrease by one-half of its initial concentration.
Time Frame: pre-dose, 0.5, 1, 2, 4, 6, 24, 48, 72 and 96 hours post dose on Day 1
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Dose Escalation: Enzalutamide 80 mg | Dose Escalation: Enzalutamide 160 mg
Number analyzed (Participants) | 7 | 8
hours | 280 (170) | 198 (105)

13. Primary Outcome: Dose Escalation Phase: Apparent Oral Clearance (CL/F) of Enzalutamide After Single Dosing
Description: Apparent oral clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. It was obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed.
Time Frame: pre-dose, 0.5, 1, 2, 4, 6, 24, 48, 72 and 96 hours post dose on Day 1
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: liter per hour
Arm/Group | Dose Escalation: Enzalutamide 80 mg | Dose Escalation: Enzalutamide 160 mg
Number analyzed (Participants) | 7 | 8
liter per hour | 0.426 (0.160) | 0.382 (0.115)

14. Primary Outcome: Dose Escalation Phase: Apparent Volume of Distribution (Vz/F) of Enzalutamide After Single Dosing
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed.
Time Frame: pre-dose, 0.5, 1, 2, 4, 6, 24, 48, 72 and 96 hours post dose on Day 1
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: liter
Arm/Group | Dose Escalation: Enzalutamide 80 mg | Dose Escalation: Enzalutamide 160 mg
Number analyzed (Participants) | 7 | 8
liter | 151 (73.6) | 94.5 (13.7)

15. Primary Outcome: Dose-Escalation Phase: Maximum Plasma Concentration (Cmax) of Enzalutamide and Its Metabolites After Multiple Dosing
Description: Carboxylic Acid (M1) and N-desmethyl (M2) are two metabolites of Enzalutamide.
Time Frame: pre-dose, 0.5, 1, 2, 4, 6, and 24 hours post-dose on Day 50
Population: PK analysis population included all participants who had at least 1 dose of Enzalutamide and had sufficient PK data to calculate at least 1 of the PK parameters of interest in at least 1 treatment period. Here, number of participants analyzed signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: micrograms per milliliter
Arm/Group | Dose Escalation: Enzalutamide 80 mg | Dose Escalation: Enzalutamide 160 mg
Number analyzed (Participants) | 3 | 6
micrograms per milliliter
  Enzalutamide | 11.6 (1.95) | 15.3 (2.62)
  M1 | 1.77 (0.521) | 6.24 (2.28)
  M2 | 6.42 (0.132) | 14.1 (3.66)

16. Primary Outcome: Dose-Escalation Phase: Time to Reach Maximum Plasma Concentration (Tmax) of Enzalutamide and Its Metabolites After Multiple Dosing
Description: Carboxylic Acid (M1) and N-desmethyl (M2) are two metabolites of Enzalutamide.
Time Frame: pre-dose, 0.5, 1, 2, 4, 6, and 24 hours post-dose on Day 50
Population: as for outcome 15
Measure: Median (Full Range); unit: hours
Arm/Group | Dose Escalation: Enzalutamide 80 mg | Dose Escalation: Enzalutamide 160 mg
Number analyzed (Participants) | 3 | 6
hours
  Enzalutamide | 0.500 [0.00 to 5.50] | 1.00 [0.570 to 4.00]
  M1 | 5.70 [0.500 to 24.0] | 2.29 [0.00 to 24.0]
  M2 | 24.0 [0.570 to 24.0] | 0.58 [0.00 to 24.0]

17. Primary Outcome: Dose-Escalation Phase: Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau) of Enzalutamide and Its Metabolites After Multiple Dosing
Description: Area under the plasma concentration versus time-curve from time zero to end of dosing interval (AUCtau), where dosing interval was 24 hours. Carboxylic Acid (M1) and N-desmethyl (M2) are two metabolites of Enzalutamide.
Time Frame: pre-dose, 0.5, 1, 2, 4, 6, and 24 hours post-dose on Day 50
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: milligram*hour per milliliter
Arm/Group | Dose Escalation: Enzalutamide 80 mg | Dose Escalation: Enzalutamide 160 mg
Number analyzed (Participants) | 3 | 6
milligram*hour per milliliter
  Enzalutamide | 207 (24.3) | 325 (61.6)
  M1 | 33.0 (13.0) | 120 (56.0)
  M2 | 140 (6.08) | 317 (89.4)

18. Primary Outcome: Dose-Escalation Phase: Apparent Oral Clearance (CL/F) of Enzalutamide After Multiple Dosing
Description: as for outcome 13
Time Frame: pre-dose, 0.5, 1, 2, 4, 6, and 24 hours post-dose on Day 50
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: liter per hour
Arm/Group | Dose Escalation: Enzalutamide 80 mg | Dose Escalation: Enzalutamide 160 mg
Number analyzed (Participants) | 3 | 6
liter per hour | 0.390 (0.0491) | 0.507 (0.0906)

19. Primary Outcome: Dose-Escalation Phase: Peak-to-Trough Ratio of Enzalutamide and Its Metabolites After Multiple Dosing
Description: Peak-to-trough ratio was calculated by dividing Cmax with Cmin of Enzalutamide and its Metabolites. Carboxylic Acid (M1) and N-desmethyl (M2) are two metabolites of Enzalutamide. Cmax was maximum plasma concentration during the dosing interval and Cmin was minimum observed plasma concentration during the dosing interval.
Time Frame: pre-dose, 0.5, 1, 2, 4, 6, and 24 hours post-dose on Day 50
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Dose Escalation: Enzalutamide 80 mg | Dose Escalation: Enzalutamide 160 mg
Number analyzed (Participants) | 3 | 6
ratio
  Enzalutamide | 1.39 (0.400) | 1.14 (0.174)
  M1 | 1.32 (0.407) | 1.42 (0.388)
  M2 | 0.999 (0.0012) | 1.00 (0.0420)

20. Primary Outcome: Dose-Escalation Phase: Accumulation Ratio of AUC24 of Enzalutamide and Its Metabolites After Multiple Dosing
Description: Accumulation Ratio was defined as the ratio of AUC24 of Day 50 to AUC24 of Day 1, where AUC24 was area under the plasma concentration-time curve from time zero to 24 hours post-dose. Carboxylic Acid (M1) and N-desmethyl (M2) are two metabolites of Enzalutamide.
Time Frame: pre-dose, 0.5, 1, 2, 4, 6, and 24 hours post-dose on Day 1 and 50
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Dose Escalation: Enzalutamide 80 mg | Dose Escalation: Enzalutamide 160 mg
Number analyzed (Participants) | 3 | 6
ratio
  Enzalutamide | 17.9 (2.69) | 9.39 (3.75)
  M1 | 47.6 (21.4) | 68.0 (35.8)
  M2 | 157 (48.2) | 77.8 (35.7)

21. Secondary Outcome: Dose-Expansion Phase: Trough Plasma Concentration for Enzalutamide
Time Frame: pre-dose on Day 57
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: micrograms per milliliter
Groups:
- Dose Expansion: Enzalutamide 160 mg + Anastrozole 1 mg; Dose Expansion: Enzalutamide 160 mg + Exemestane 25 mg: Participants received enzalutamide 160 mg (four 40 mg) capsule in combination with the exemestane 25 mg tablet, orally, once daily until documented disease progression, initiation of a new antitumor treatment, an intolerable adverse event (including any seizure), noncompliance, withdrawal of consent, discontinuation by sponsor, or investigator. Participants were followed-up until 30 days after last dose of study drug or before initiation of a new antitumor or investigational therapy, whichever occurred first.
Arm/Group | Dose Expansion: Enzalutamide 160 mg | Dose Expansion: Enzalutamide 160 mg + Anastrozole 1 mg | Dose Expansion: Enzalutamide 160 mg + Exemestane 25 mg | Dose Expansion: Enzalutamide 160 mg + Exemestane 50 mg | Dose Expansion: Enzalutamide 160 mg + Fulvestrant 500 mg
Number analyzed (Participants) | 3 | 9 | 5 | 12 | 7
micrograms per milliliter | 13.40 (2.51) | 14.33 (3.99) | 13.52 (2.62) | 12.41 (3.76) | 11.62 (4.69)

ADVERSE EVENTS:
Time Frame: Day 1 up to 30 days after the last dose of study drug or before initiation of a new systemic antitumor treatment, whichever occurred first (up to 3.5 years)
Description: Same event may appear as both an AE and SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event.
Arm/Group | Dose Escalation: Enzalutamide 80 mg | Dose Escalation: Enzalutamide 160 mg | Dose Expansion: Enzalutamide 160 mg | Dose Expansion: Enzalutamide 160 mg + Anastrozole 1 mg | Dose Expansion: Enzalutamide 160 mg + Exemestane 25 mg | Dose Expansion: Enzalutamide 160 mg + Exemestane 50 mg | Dose Expansion: Enzalutamide 160 mg + Fulvestrant 500 mg
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/8 | 1/14 | 0/20 | 0/16 | 0/23 | 0/11
Serious Adverse Events (participants affected / at risk) | 2/7 | 1/8 | 2/14 | 1/20 | 5/16 | 3/23 | 2/11
Other Adverse Events (participants affected / at risk) | 7/7 | 8/8 | 14/14 | 20/20 | 15/16 | 21/23 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Escalation: Enzalutamide 80 mg (N=7) | Dose Escalation: Enzalutamide 160 mg (N=8) | Dose Expansion: Enzalutamide 160 mg (N=14) | Dose Expansion: Enzalutamide 160 mg + Anastrozole 1 mg (N=20) | Dose Expansion: Enzalutamide 160 mg + Exemestane 25 mg (N=16) | Dose Expansion: Enzalutamide 160 mg + Exemestane 50 mg (N=23) | Dose Expansion: Enzalutamide 160 mg + Fulvestrant 500 mg (N=11)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pericardial Effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Adrenal Insufficiency (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastritis Erosive (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
In-Stent Coronary Artery Restenosis (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Humerus Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tumour Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Obstructive Uropathy (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Renal Failure Acute (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ureteric Obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Escalation: Enzalutamide 80 mg (N=7) | Dose Escalation: Enzalutamide 160 mg (N=8) | Dose Expansion: Enzalutamide 160 mg (N=14) | Dose Expansion: Enzalutamide 160 mg + Anastrozole 1 mg (N=20) | Dose Expansion: Enzalutamide 160 mg + Exemestane 25 mg (N=16) | Dose Expansion: Enzalutamide 160 mg + Exemestane 50 mg (N=23) | Dose Expansion: Enzalutamide 160 mg + Fulvestrant 500 mg (N=11)
Anaemia (Blood and lymphatic system disorders) | 2 | 2 | 1 | 1 | 5 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 2 | 0 | 1 | 1
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lymph Node Pain (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 1
Palpitations (Cardiac disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Angina Pectoris (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Cardiac Tamponade (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dry Eye (Eye disorders) | 0 | 2 | 0 | 1 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Eye Movement Disorder (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eyelid Oedema (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lacrimation Increased (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abnormal Sensation In Eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vision Blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Visual Acuity Reduced (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 5 | 3 | 2 | 7 | 3
Diarrhoea (Gastrointestinal disorders) | 3 | 1 | 2 | 6 | 4 | 3 | 4
Constipation (Gastrointestinal disorders) | 0 | 2 | 2 | 3 | 3 | 3 | 3
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 0 | 4 | 0 | 2 | 2 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 0 | 3 | 1 | 0 | 2 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 2 | 1 | 1 | 0 | 2
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal Distension (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 1
Dry Mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 0
Epigastric Discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eructation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal Pain Lower (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1
Frequent Bowel Movements (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 2 | 8 | 12 | 8 | 12 | 8
Chills (General disorders) | 0 | 1 | 1 | 2 | 0 | 0 | 0
Oedema Peripheral (General disorders) | 0 | 0 | 2 | 1 | 1 | 1 | 1
Pyrexia (General disorders) | 0 | 1 | 1 | 1 | 0 | 2 | 1
Asthenia (General disorders) | 0 | 0 | 1 | 5 | 0 | 1 | 0
Axillary Pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chest Discomfort (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Early Satiety (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Gait Disturbance (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Influenza Like Illness (General disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 0
Irritability (General disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Spinal Pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Suprapubic Pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Local Swelling (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hepatomegaly (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Drug Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Breast Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 1 | 0
Cystitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ear Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Infected Cyst (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia Bacterial (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 1
Skin Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 2 | 1
Viral Upper Respiratory Tract (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Acute Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Herpes Zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Open Wound (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 2 | 2
Aspartate Aminotransferase Increased (Investigations) | 4 | 1 | 0 | 2 | 1 | 0 | 0
Alanine Aminotransferase Increased (Investigations) | 2 | 0 | 0 | 1 | 2 | 0 | 0
Blood Alkaline Phosphatase Increased (Investigations) | 1 | 2 | 0 | 0 | 2 | 1 | 1
International Normalised Ratio Increased (Investigations) | 2 | 0 | 0 | 0 | 1 | 0 | 0
Weight Decreased (Investigations) | 0 | 2 | 0 | 3 | 4 | 1 | 3
Blood Lactate Dehydrogenase Increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lymphocyte Count Decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
White Blood Cell Count Decreased (Investigations) | 0 | 1 | 0 | 2 | 3 | 1 | 0
Activated Partial Thromboplastin Time Prolonged (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Blood Bilirubin Increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 1 | 0
Neutrophil Count Decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Platelet Count Decreased (Investigations) | 0 | 0 | 0 | 0 | 2 | 1 | 0
Malignant Pleural Effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Skin Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tumour Associated Fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tumour Haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Metastases To Ovary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Breast Pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Vulvovaginal Dryness (Reproductive system and breast disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0
Ovarian Cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 1 | 4 | 1 | 1 | 0 | 5 | 2
Hot Flush (Vascular disorders) | 0 | 0 | 4 | 5 | 2 | 4 | 3
Lymphoedema (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Device Related Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 3 | 0 | 1 | 3 | 2 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 1 | 1 | 1 | 10 | 5 | 4 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 1 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 1 | 1 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 2 | 2 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1
Increased Appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Iron Deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 2 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0
Micturition Urgency (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Renal Failure Acute (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Urinary Incontinence (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 2 | 3 | 3 | 4 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 4 | 2 | 2 | 2 | 4
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 2 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 1 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Upper-Airway Cough Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 2 | 1 | 2 | 1
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 2 | 2 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 2 | 0 | 2
Blood Blister (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 3 | 0
Rash Generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Night Sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 1 | 2 | 2 | 6 | 3
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 5 | 3 | 2 | 5 | 6
Groin Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 3 | 1 | 4 | 0
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Joint Stiffness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 2 | 1 | 1 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 3 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 1
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2 | 2 | 1 | 2
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 2 | 2 | 1 | 0
Pain In Jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 2 | 2
Dizziness (Nervous system disorders) | 2 | 1 | 3 | 2 | 3 | 2 | 3
Headache (Nervous system disorders) | 1 | 1 | 3 | 3 | 1 | 2 | 4
Neuropathy Peripheral (Nervous system disorders) | 1 | 2 | 0 | 2 | 1 | 0 | 0
Cognitive Disorder (Nervous system disorders) | 0 | 0 | 2 | 1 | 3 | 0 | 4
Memory Impairment (Nervous system disorders) | 0 | 0 | 2 | 2 | 0 | 2 | 1
Restless Legs Syndrome (Nervous system disorders) | 1 | 1 | 0 | 2 | 0 | 1 | 2
Disturbance In Attention (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Sciatica (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 4 | 1 | 0 | 2
Peripheral Sensory Neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sinus Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 3 | 1 | 3 | 2 | 1 | 2
Insomnia (Psychiatric disorders) | 0 | 2 | 1 | 5 | 2 | 2 | 1
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0 | 1 | 2 | 2
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 3
Confusional State (Psychiatric disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0
Hallucination, Visual (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 3 | 8 | 9 | 7 | 12 | 8
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Faecal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
Prioritization of outcome measures as primary and secondary was based on the study team's discretion.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.